CLINICAL TRIAL: NCT03595059
Title: A Phase 1 First-in-Human Study With ABBV-155 Alone and in Combination With Taxane Therapy in Adults With Relapsed and/or Refractory Solid Tumors
Brief Title: A Study With ABBV-155 Alone and in Combination With Taxane Therapy in Adults With Relapsed and/or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M16-573; 2020-002495-12 (EudraCT Number)
Record Dates: First submitted 2018-07-12; First posted 2018-07-23 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors
Keywords: Cancer; Advanced Solid Tumors; Relapsed and/or Refractory Solid Tumors; ABBV-155; Taxane; Paclitaxel; Docetaxel; breast cancer; non-small cell lung cancer (NSCLC); small cell lung cancer (SCLC)
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Paclitaxel; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Escalation 1a: ABBV-155 (Experimental): Participants will be administered ABBV-155 (various doses).
  Interventions: Drug: ABBV-155
- Escalation 1b: ABBV-155 + paclitaxel or docetaxel (Experimental): Participants will be administered ABBV-155 (various doses) in combination with paclitaxel or docetaxel .
  Interventions: Drug: ABBV-155; Drug: Paclitaxel; Drug: Docetaxel
- Expansion 2a: ABBV-155 in SCLC (Experimental): Description: Participants with small cell lung cancer (SCLC) will administer ABBV-155 (at the recommended Phase 2 dose).
  Interventions: Drug: ABBV-155
- Expansion 2b: ABBV-155 + paclitaxel in Breast Cancer (Experimental): Participants with breast cancer will be administered ABBV-155 (at the recommended Phase 2 dose identified for combination with paclitaxel in part 1b) in combination with paclitaxel.
  Interventions: Drug: ABBV-155; Drug: Paclitaxel
- Expansion 2b: ABBV-155 + docetaxel in NSCLC (Experimental): Participants with non-small cell lung cancer (NSCLC) will be administered ABBV-155 (at or near the recommended Phase 2 dose identified for combination with paclitaxel in part 1b) in combination with docetaxel.
  Interventions: Drug: ABBV-155; Drug: Docetaxel

INTERVENTIONS:
Drug: ABBV-155 — Intravenous (IV) Infusion
Drug: Paclitaxel — Intravenous (IV) Infusion
  Arms: Escalation 1b: ABBV-155 + paclitaxel or docetaxel; Expansion 2b: ABBV-155 + paclitaxel in Breast Cancer
Drug: Docetaxel — Intravenous (IV) Infusion
  Arms: Escalation 1b: ABBV-155 + paclitaxel or docetaxel; Expansion 2b: ABBV-155 + docetaxel in NSCLC

SUMMARY:
An open-label, dose-escalation (Part 1), dose-expansion (Part 2) study to assess the safety, pharmacokinetics (PK), and preliminary efficacy of ABBV-155 alone and in combination with paclitaxel or docetaxel.

In Part 1 (dose escalation), participants will receive escalating doses of ABBV-155 monotherapy (Part 1a) or ABBV-155 in combination with paclitaxel or docetaxel (Part 1b).

In Part 2 (dose expansion), participants will receive ABBV-155 monotherapy or in combination therapy. The ABBV-155 monotherapy cohort will enroll participants with relapsed or refractory (R/R) small cell lung cancer (SCLC) (Part 2a); the ABBV-155 plus a taxane (paclitaxel or docetaxel) combination cohort will enroll participants with R/R non-small cell lung cancer (NSCLC) and breast cancer (Part 2b).

DETAILED DESCRIPTION:
The Escalation cohorts (Part 1) have been completed. The expansion cohorts (Part 2) are open to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologic or cytologic diagnosis of a malignant solid tumor.
* Participants enrolled in Part 2a (monotherapy, dose expansion) must have small cell lung cancer (SCLC) diagnosis; participants enrolled to Part 2b (combination therapy, dose expansion) must have either NSCLC or HR-positive/HER2-negative breast cancer.
* Measurable disease defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* An Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
* Failure of at least 1 prior systemic chemotherapy including all available standard therapies for participants in the dose-escalation phase (Parts 1a and 1b) including the safety lead-in phase (Japan only).
* All participants with breast cancer for subjects in the dose-expansion phase (Part 2b only) must have the following:

  * Locally advanced or metastatic HR-positive/HER2-negative breast cancer after failing cyclin-dependent kinase (CDK)4/6 inhibitor-based therapy.
  * HR-positivity and HER-2-negativity should be confirmed based on American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) criteria.
* All participants with non-small cell lung cancer (NSCLC) for participants in the dose-expansion phase (Part 2b only) must have R/R NSCLC after at least 1 line of therapy. Participants with activating mutations in EGFR, ALK/ROS1, BRAF genes, or with positive expression of PD-L1 must have been treated with the appropriate targeted therapies.
* All participants with SCLC in the dose-expansion phase (Part 2a only) must have R/R SCLC from at least 1 line of therapy which includes a platinum-based therapy with or without an anti-PD-1/PD-L1 therapy.
* All participants with either breast cancer or NSCLC must have the following if exposed to prior taxane-based therapy:

  * No history of taxane allergy (Part 1b and Part 2b only).
  * Disease that has relapsed or progressed at least 2 months after most recent exposure to any taxane-based therapy.
* Available tumor tissue suitable for immunohistochemistry testing.
* Adequate kidney, liver, and hematologic laboratory values as described in the protocol.

Exclusion Criteria:

* Untreated brain or meningeal metastases (participants with a history of metastases may be eligible based on details described in the protocol).
* Grade 2 or higher peripheral neuropathy (only applies to participants who would receive taxane therapy).
* Unresolved Grade 2 or higher toxicities related to previous anticancer therapy except alopecia.
* Known active infection of hepatitis B, hepatitis C, or human immunodeficiency virus with exceptions as described in the protocol.
* Recent history (within 6 months) of congestive heart failure (defined in the protocol), ischemic cardiovascular event, cardiac arrhythmia requiring pharmacological or surgical intervention, pericardial effusion, or pericarditis.
* Any history of hypersensitivity to any ingredients of ABBV-155 will be excluded. For combination therapy only (Parts 1b and 2b), no history of serious allergic reaction to any taxane or any ingredients used in taxane formulation (e.g., cremaphor).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
MTD and/or RPTD of ABBV-155 | Up to approximately 21 days after initial dose of study drug
  The Maximum Tolerated Dose (MTD) and/or the Recommended Phase Two Dose (RPTD) of ABBV-155 will be determined during the dose escalation phase (Part 1).
Overall Response Rate (ORR) | Up to approximately 2 to 6 months
  ORR is defined as the percentage of participants with documented best response partial response (PR) or better according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AE) | Up to approximately 12 months
  An AE is defined as any untoward medical occurrence in a subject or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Duration of Response (DOR) | Up to approximately 12 months
  DOR is defined as the number of days from the date of first documented response (PR or better) to the date of the first documented disease progression (PD) or death due to disease, whichever occurs first.
Rate of Complete Response (CR) | Up to approximately 2 to 6 months
  CR is defined as the percentage of participants with documented best response CR according to RECIST version 1.1
Progression-Free Survival (PFS) | Up to approximately 12 months
  PFS is defined as the number of days from the date of first dose of study drug to the date of the first documented PD or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 12 months after last dose of study drug
  OS is defined as the number of days from the date of first study drug to the date of death due to any cause.
Cmax of ABBV-155 | Up to approximately 48 days
  Maximum plasma concentration (Cmax).
Tmax of ABBV-155 | Up to approximately 48 days
  Time to maximum plasma concentration (Tmax).
Terminal Phase Elimination Rate constant of ABBV-155 | Up to approximately 48 days
  Terminal phase elimination rate constant of ABBV-155
AUCt of ABBV-155 | Up to approximately 48 days
  Area under the plasma concentration versus time curve (AUC) from time 0 to the time of the last measurable concentration (AUCt).
AUCinf of ABBV-155 | Up to approximately 48 days
  AUC from time 0 to infinite time (AUCinf).
QTcF Change from Baseline | Up to approximately 8 days
  QT interval measurement corrected by Fridericia's formula (QTcF) mean change from baseline by dose level of ABBV-155 Monotherapy.
t1/2 of ABBV-155 | Up to approximately 48 days
  Terminal elimination half-life (t1/2).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (40):
- United States (21):
  - University of Alabama at Birmingham - Main /ID# 214024, Birmingham, Alabama
  - Highlands Oncology Group, PA /ID# 201568, Springdale, Arkansas
  - UC Irvine Medical Center - Chao Family Comprehensive Cancer Center /ID# 206105, Orange, California
  - Duplicate_Cedars-Sinai Medical Center-West Hollywood /ID# 204267, West Hollywood, California
  - Univ of Colorado Cancer Center /ID# 208365, Aurora, Colorado
  - Yale University, Yale Cancer Center /ID# 201542, New Haven, Connecticut
  - AdventHealth Orlando /ID# 227242, Orlando, Florida
  - Northwestern University Feinberg School of Medicine /ID# 201563, Chicago, Illinois
  - Duplicate_Johns Hopkins Bayview Med Cnt /ID# 215095, Baltimore, Maryland
  - Johns Hopkins Hospital /ID# 201320, Baltimore, Maryland
  - Dana-Farber Cancer Institute /ID# 201564, Boston, Massachusetts
  - Duplicate_Henry Ford Hospital /ID# 226852, Detroit, Michigan
  - Northwell Health - Marcus Ave /ID# 204376, New Hyde Park, New York
  - Carolina BioOncology Institute /ID# 201577, Huntersville, North Carolina
  - Univ Hosp Cleveland /ID# 201567, Cleveland, Ohio
  - University of Oklahoma, Stephenson Cancer Center /ID# 206820, Oklahoma City, Oklahoma
  - Lifespan Cancer Institute at Rhode Island Hospital /ID# 204256, Providence, Rhode Island
  - Vanderbilt Ingram Cancer Center /ID# 201575, Nashville, Tennessee
  - Mary Crowley Cancer Research /ID# 214168, Dallas, Texas
  - MD Anderson Cancer Center /ID# 201558, Houston, Texas
  - NEXT Oncology /ID# 204893, San Antonio, Texas
- Peter MacCallum Cancer Center /ID# 241676, Melbourne, New South Wales, Australia
- Canada (2):
  - Duplicate_Cross Cancer Institute /ID# 213838, Edmonton, Alberta
  - University Health Network_Princess Margaret Cancer Centre /ID# 204539, Toronto, Ontario
- Israel (2):
  - The Chaim Sheba Medical Center /ID# 230812, Ramat Gan, Tel Aviv
  - Rambam Health Care Campus /ID# 230813, Haifa
- Japan (2):
  - National Cancer Center Hospital East /ID# 215130, Kashiwa-shi, Chiba
  - National Cancer Center Hospital /ID# 215003, Chuo-ku, Tokyo
- Netherlands (4):
  - Maastricht Universitair Medisch Centrum /ID# 225220, Maastricht, Limburg
  - Antoni van Leeuwenhoek /ID# 222260, Amsterdam, North Holland
  - Erasmus Medisch Centrum /ID# 222341, Rotterdam, South Holland
  - Universitair Medisch Centrum Utrecht /ID# 222357, Utrecht
- Pan American Center for Oncology Trials, LLC /ID# 232128, Rio Piedras, Puerto Rico
- South Korea (2):
  - National Cancer Center /ID# 241095, Goyang-si, Gyeonggido
  - Yonsei University Health System Severance Hospital /ID# 240648, Seoul
- Spain (2):
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 239997, Madrid
  - Hospital Universitario 12 de Octubre /ID# 239999, Madrid
- Taiwan (3):
  - National Taiwan University Hospital /ID# 205673, Taipei City, Taipei
  - China Medical University Hospital /ID# 214062, Taichung
  - National Cheng Kung University Hospital /ID# 206304, Tainan

IPD SHARING:
Plan to Share IPD: No